CLINICAL TRIAL: NCT04955431
Title: The Effects of Circadian Rhythm Disruption on the Inflammatory Response to Particulate Matter Exposure From Woodsmoke
Brief Title: Circadian Rhythm Disruption Effects on Smoke Inhalation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, John Quindry, Professor and Chair, University of Montana
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB# is 83-21
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Inflammation; Sleep Deprivation; Circadian Rhythm Sleep Disorder, Shift Work Type; Smoke Inhalation
MeSH Terms: conditions — Inflammation; Sleep Deprivation; Sleep Disorders, Circadian Rhythm; Smoke Inhalation Injury

STUDY DESIGN:
Intervention Model Description: Randomized cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Sleep (with 250 ug/m^3 PM2.5) (Placebo Comparator): Participants will have a normal sleep opportunity the night prior to reporting to the lab for the simulated firefighting session (250 ug/m^3 PM2.5 with moderate intensity exercise).
  Interventions: Behavioral: Normal Sleep
- Restricted Sleep (with 250 ug/m^3 PM2.5) (Experimental): Participants will have a restricted sleep opportunity (~4 hours) the night prior to reporting to the lab for the simulated firefighting session (250 ug/m^3 PM2.5 with moderate intensity exercise).
  Interventions: Behavioral: Sleep Restriction

INTERVENTIONS:
Behavioral: Sleep Restriction — Participants will be allowed ~4 hour sleep opportunity during the restricted night of sleep prior to reporting to lab for a simulated firefighting session.
  Other Names: Circadian Rhythm Disruption; SR
  Arms: Restricted Sleep (with 250 ug/m^3 PM2.5)
Behavioral: Normal Sleep — Participants will be allowed ~8 hour sleep opportunity the night of sleep prior to reporting to lab for a simulated firefighting session.
  Other Names: NS
  Arms: Normal Sleep (with 250 ug/m^3 PM2.5)

SUMMARY:
Particulate matter exposure during smoke inhalation provokes inflammatory immune responses in people exposed to burning biomass including fire fighters and civilians. Persistent occupational exposure to particulate matter represents a unique hazard for firefighters, underpinning a burgeoning research area. This trial will evaluate the effects of sleep deprivation and circadian rhythm disruption on the inflammatory response to woodsmoke associated particulate matter exposure. Participants will undergo 2 experimental trials in a randomized cross-over design. Participants will have either an 8-hour sleep opportunity or a 4-hour sleep opportunity prior to reporting to lab for a 45 minute simulated firefighting trial (wood smoke associated particulate matter filtered to 2.5 um at a concentration of 250 ug/m^3, while exercising at a moderate intensity). The effects of sleep restriction and simulated firefighting will be measured.

DETAILED DESCRIPTION:
Participants: Healthy college age males (n = 15), free from disordered sleep and without recent trans-meridian travel (within the last 2 weeks) will be recruited for this study. Participants will complete chronotype questionnaires (Morningness-Eveningness Questionnaire; MEQ, Munich Chronotype Questionnaire; MCTQ) to establish intermediate chronotypes. This will minimize the effect of circadian preference on the morning exposure to smoke. Participants will subsequently be outfitted with activity monitors (ActiCal) to monitor sleep and physical activity throughout the experimental duration. Participants will be asked to maintain a normal sleep schedule for at least 3 days leading up to the experimental trials and keep a sleep log to verify.

Experimental Trials: Participants will undergo 2 experimental trials in a randomized cross-over design, with at least 1 week washout period between trials; 1) NS-250: Normal Sleep with exposure to woodsmoke at 250 µg/m^3, and RS-250: Restricted Sleep with exposure to woodsmoke at 250 µg/m^3. Participants will have an 8-hour sleep opportunity in their own home during the NS trials (22:00-06:00), and a 4-hour sleep opportunity during the RS trials (00:00-04:00). In all trials, participants will report to the laboratory at 07:30 the morning after the experimental sleep night. PM exposure will occur from 08:00-08:45 while cycling at 70% heart rate reserve (HRR) to simulate the physical demands of firefighting.

Exhaled Breath Condensate (EBC): EBC will be collected using standardized 10 minute collection techniques. In order to preserve sample integrity for potentially labile biomarkers (e.g., oxidative stress), sample pH will be measured immediately prior to aliquoting in multiple cryotubes (500-700µl), flash freezing, and storage at -80 degrees C until further assay. Standardized biomarker panels for oxidative stress and inflammation will be performed using a single thaw approach.

Inflammatory biomarker analysis: Blood will be collected into heparinized vacutainers before (PRE) and immediately following (POST) PM2.5 exposure and spun down for plasma collection. Plasma will be assayed for inflammatory biomarkers (interleukin (IL)-6, tumor necrosis factor (TNF)-α, pentraxin-3, and C-reactive protein (CRP)) using standard enzyme linked immunosorbent assays (ELISA).

Circadian Rhythm Assessment: Throughout the experimental protocol, circadian rhythms will be assessed in two ways; 1) Actigraphy and 2) Clock gene expression in buccal cell swabs. Acticals will be worn throughout to gather sleep variables (timing, duration, quality). Clock gene expression (CLOCK, BMAL1, PER2) will be measured in swabs taken from the cheek at 6 hour intervals (00:00, 06:00, 12:00, 18:00) to assess the effects of sleep deprivation on the molecular circadian rhythm. Cheek swabs will be immediately placed in RNA stabilization buffer until isolation. Swabs taken at 00:00 will be performed with minimal exposure to light to avoid disruption of sleep. These methods have been used previously to assess normal and disrupted sleep.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* 18 - 44 years of age

Exclusion Criteria:

* Preexisting cardiometabolic and/or pulmonary diseases
* Preexisting sleep disorder
* Smoking (current or within last year)

Ages: 18 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Quindry, PhD, Principal Investigator — University of Montana
Locations (1):
- School of Integrative Physiology and Athletic Training, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. Blinded anonymized outcomes data will be shared via publication and presentation of results.

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Sleep (With 250 ug/m^3 PM2.5) Then Restricted Sleep (With 250 ug/m^3 PM2.5): Participants will complete two sessions in the lab. During their first session, they will have a normal sleep opportunity the night prior to reporting to the lab for the simulated firefighting session (250 ug/m^3 PM2.5 with moderate intensity exercise).
  Normal Sleep: Participants will be allowed ~8 hour sleep opportunity the night of sleep prior to reporting to lab for a simulated firefighting session.
  During their second session, participants will have a restricted sleep opportunity (~4 hours) the night prior to reporting to the lab for the simulated firefighting session (250 ug/m^3 PM2.5 with moderate intensity exercise).
  Sleep Restriction: Participants will be allowed ~4 hour sleep opportunity during the restricted night of sleep prior to reporting to lab for a simulated firefighting session.
- Restricted Sleep (With 250 ug/m^3 PM2.5) Then Normal Sleep (With 250 ug/m^3 PM2.5): Participants will complete two sessions in the lab. During their first session, participants will have a restricted sleep opportunity (~4 hours) the night prior to reporting to the lab for the simulated firefighting session (250 ug/m^3 PM2.5 with moderate intensity exercise).
  Sleep Restriction: Participants will be allowed ~4 hour sleep opportunity during the restricted night of sleep prior to reporting to lab for a simulated firefighting session.
  During their second session, participants will have a normal sleep opportunity the night prior to reporting to the lab for the simulated firefighting session (250 ug/m^3 PM2.5 with moderate intensity exercise).
  Normal Sleep: Participants will be allowed ~8 hour sleep opportunity the night of sleep prior to reporting to lab for a simulated firefighting session.
Period: Overall Study
Arm/Group | Normal Sleep (With 250 ug/m^3 PM2.5) Then Restricted Sleep (With 250 ug/m^3 PM2.5) | Restricted Sleep (With 250 ug/m^3 PM2.5) Then Normal Sleep (With 250 ug/m^3 PM2.5)
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Sleep (With 250 ug/m^3 PM2.5) Then Restricted Sleep (With 250 ug/m^3 PM2.5) | Restricted Sleep (With 250 ug/m^3 PM2.5) Then Normal Sleep (With 250 ug/m^3 PM2.5) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (3.56) | 25.0 (5.0) | 24.4 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Blood IL-6 [Mean (Standard Deviation); unit: pg/mL] — Baseline interleukin-6 (IL-6) levels were determined from blood samples taken before interventions.
  pg/mL | 0.69 (0.31) | 0.80 (0.79) | 0.75 (0.59)

OUTCOME MEASURES:

1. Primary Outcome: Blood Inflammation
Description: IL-6 will be measured in the plasma
Time Frame: samples collected at baseline, immediately post exposure
Population: Blood plasma was used to measure IL-6 using a commercially available ELISA.
Measure: Mean (Standard Error); unit: pg/mL
Units Other Than Participants: Plasma
Arm/Group | Normal Sleep (With 250 ug/m^3 PM2.5) | Restricted Sleep (With 250 ug/m^3 PM2.5)
Number analyzed (Participants) | 10 | 10
Number analyzed (Plasma) | 20 | 20
pg/mL
  Baseline | 0.69 (0.10) | 0.79 (0.25)
  POST | 2.33 (0.33) | 1.63 (0.25)
Statistical Analysis 1: Comparison: Normal Sleep (With 250 ug/m^3 PM2.5) vs Restricted Sleep (With 250 ug/m^3 PM2.5); Test type: Other — We performed a 2-way Repeated Measures ANOVA to compare changes in blood IL-6 levels from baseline to post simulated firefighting on control days (Normal Sleep) and experimental days (Sleep Restriction); p < 0.05, ANOVA

2. Secondary Outcome: Exhaled Breath Condensate Pentraxin-3
Description: Pentraxin-3 will be measured in EBC of participants at baseline (PRE) and after exercise (POST) on two trial days. One trial day will be after a normal night of sleep (Normal Sleep) and the other trial will be after sleep restriction to 4 hours (Restricted Sleep). The value is determined through ELISA method, represented in ng/mL, where higher levels indicate worse response.
Time Frame: samples collected at baseline, immediately post exposure
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Sleep (With 250 ug/m^3 PM2.5) | Restricted Sleep (With 250 ug/m^3 PM2.5)
Number analyzed (Participants) | 10 | 10
ng/mL
  PRE | 0.97 (0.04) | 0.95 (0.02)
  POST | 0.96 (0.02) | 0.96 (0.03)
Statistical Analysis 1: Comparison: Normal Sleep (With 250 ug/m^3 PM2.5); Test type: Other — RM-ANOVA; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout participation in the study, which was roughly three weeks per participant.
Description: The experimental interventions used in this study (mild smoke inhalation, moderate intensity exercise, mild sleep restriction) were not of a life threatening nature and our participants were healthy. As such, none of our participants were at risk for All-Cause Mortality.
Arm/Group | Normal Sleep (With 250 ug/m^3 PM2.5) | Restricted Sleep (With 250 ug/m^3 PM2.5)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Our study was limited by a smaller sample size than we had anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT04955431/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT04955431/SAP_001.pdf